CLINICAL TRIAL: NCT02976220
Title: Health Outcomes Patient Education
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Cricket Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-19626
Record Dates: First submitted 2016-09-28; First posted 2016-11-29 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digital Education (Experimental): 1 month digital education program
  Interventions: Other: Digital Education

INTERVENTIONS:
Other: Digital Education — Online videos, illustrations, and text materials designed to improve participants' awareness and understanding of kidney function, kidney disease, kidney failure options, peritoneal dialysis, home hemodialysis, in-center hemodialysis, kidney transplant, medical management, and treatment decision. Also includes online messaging system and discussion board designed to allow participants to message study nurse and peer mentor, as well as to engage in group discussion in an open forum and about specific scenarios.

SUMMARY:
This study is designed to evaluate the feasibility of using digital-enabled education in clinical care in order to improve patient outcomes related to end-stage renal disease (ESRD). If effective, educational interventions could be used to improve the long-term survival of patients with chronic kidney disease (CKD) and to make clinical care for these patients more cost effective.

DETAILED DESCRIPTION:
Studies have shown that educational interventions in patients nearing end-stage renal disease (ESRD) can delay the need for dialysis and increase the likelihood of the patient choosing in-home vs. in-center dialysis. Given the higher cost of in-center hemodialysis compared to in-home strategies, such as peritoneal dialysis, efforts at increasing use of in-home dialysis modalities are likely to be cost-effective. Moreover, while few studies of educational interventions have long-term follow-up, one study suggests that patients exposed to educational interventions have improved long-term survival once on dialysis.

The long-term goal is to improve clinical and patient-centered outcomes in patients transitioning from Chronic Kidney Disease Stage (CKD) IV and V to dialysis-requiring ESRD. The short-term goal of this pilot project is to evaluate the feasibility of delivering digital-enabled ESRD education to patients with CKD stage IV and V (eGFR<30ml/min/1.73m2, not yet on dialysis) in clinical care. The investigators will provide this education in the form of in-person nurse advice, online digital content including videos, and online messaging with a nurse, moderated patient group and peer mentor. The main objective of the educational program will be to 1) Increase awareness of options, 2) Prioritize options based on patient lifestyle and values, 3) Build confidence in modality decision.

The investigators will develop individualized, digitalized educational content (which includes videos, text and illustration) for patients with CKD that will increase awareness of ESRD care options including in-home hemodialysis, peritoneal dialysis and choosing not to have dialysis. Patients will enroll in a month-long program during which they have access to the educational app, including lifestyle and modality educational content and online messaging where they can access a nurse for 1 on 1 discussion, a patient mentor for 1 on 1 discussion, and a patient group for group mentorship exercises. The investigators will pilot these materials in patients at high risk of progression to dialysis and evaluate the primary outcomes of whether they were able to complete the program and make a modality choice. Secondary outcomes will include assessments to determine the intervention's impact on patient dialysis modality awareness and likelihood of choosing a home-dialysis modality. At the end of the study, the investigators will provide an insights report to the study participants' doctors and survey the doctors to ascertain their perspectives on the usefulness of the educational program for their patients' care.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 30ml/min/1.73m²
* Regular attendance at the nephrology clinic; at least two visits within the last 18 months
* Clinic notes indicate patient has had discussion with a nephrologist regarding needing dialysis in the future

Exclusion Criteria:

* Homelessness
* Non-English speaking
* No phone or no internet access on one of the following: smart phone, tablet, or computer
* No e-mail access
* Age ≥ 90 years
* Hospitalized more than twice during the last 6 months
* Dementia
* Severe cognitive impairment
* Blindness
* Deafness

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who feel ready to choose a treatment option from among home hemodialysis, in-center hemodialysis, peritoneal dialysis or conservative care | 1 month
  Number of participants who feel ready to choose a treatment option from among home hemodialysis, in-center hemodialysis, peritoneal dialysis or conservative care. Unit of measure: the change from pre- to post-educational program, # participants.

SECONDARY OUTCOMES:
General Knowledge | 1 month
  This questionnaire will include multiple choice questions designed to show if the patient gained general knowledge about kidney disease from the education program. Unit of measure: the change from pre- to post-educational program in per cent of questions each patient answered correctly.
Modality Knowledge | 1 month
  This questionnaire will include multiple choice questions designed to show if the patient understands the different options of care for end-stage renal disease, including home hemodialysis, in-center hemodialysis, peritoneal dialysis or conservative care. Unit of measure: the change from pre- to post-educational program in per cent of questions each patient answered correctly.
Self-efficacy | 1 month
  This survey consists of five questions drawn from validated surveys of self-efficacy in the chronic kidney disease population. Unit of measure: Each question is answered on a likert scale 1-5. Total score ranges from 5 to 25. Unit of measure is change in overall likert rating for each participant from pre- and post-educational program.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Dubin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center: Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Devins GM, Mendelssohn DC, Barre PE, Binik YM. Predialysis psychoeducational intervention and coping styles influence time to dialysis in chronic kidney disease. Am J Kidney Dis. 2003 Oct;42(4):693-703. doi: 10.1016/s0272-6386(03)00835-7. PMID 14520619
- [Background] Mason J, Khunti K, Stone M, Farooqi A, Carr S. Educational interventions in kidney disease care: a systematic review of randomized trials. Am J Kidney Dis. 2008 Jun;51(6):933-51. doi: 10.1053/j.ajkd.2008.01.024. Epub 2008 Apr 28. PMID 18440681
- [Background] Manns BJ, Taub K, Vanderstraeten C, Jones H, Mills C, Visser M, McLaughlin K. The impact of education on chronic kidney disease patients' plans to initiate dialysis with self-care dialysis: a randomized trial. Kidney Int. 2005 Oct;68(4):1777-83. doi: 10.1111/j.1523-1755.2005.00594.x. PMID 16164654
- [Background] U.S. Renal Data System, USRDS 2013 Annual Data Report: Atlas of Chronic Kidney Disease and End-Stage Renal Disease in the United States, National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2013.
- [Background] Devins GM, Mendelssohn DC, Barre PE, Taub K, Binik YM. Predialysis psychoeducational intervention extends survival in CKD: a 20-year follow-up. Am J Kidney Dis. 2005 Dec;46(6):1088-98. doi: 10.1053/j.ajkd.2005.08.017. PMID 16310575
- [Derived] Dubin R, Rubinsky A. A Digital Modality Decision Program for Patients With Advanced Chronic Kidney Disease. JMIR Form Res. 2019 Feb 6;3(1):e12528. doi: 10.2196/12528. PMID 30724735